CLINICAL TRIAL: NCT07141199
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of ABBV-8736 After Multiple Ascending Doses in Healthy Adult Subjects
Brief Title: A Study to Evaluate Adverse Events, How the Drug is Tolerated, and How the Drug Moves Through the Body of Intravenous Infusions of ABBV-8736 in Adult Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: M25-918
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; ABBV-8736

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1: Dose A of ABBV-8736 (Experimental): Participants will receive intravenous (IV) ABBV-8736 dose A every 2 weeks for a total of 3 doses.
  Interventions: Drug: ABBV-8736
- Group 1: Dose A of ABBV-8736 Placebo (Placebo Comparator): Participants will receive IV ABBV-8736 placebo dose A every 2 weeks for a total of 3 doses.
  Interventions: Drug: Placebo
- Group 2: Dose B of ABBV-8736 (Experimental): Participants will receive IV ABBV-8736 dose B every 2 weeks for a total of 3 doses.
  Interventions: Drug: ABBV-8736
- Group 2: Dose B of ABBV-8736 Placebo (Placebo Comparator): Participants will receive IV ABBV-8736 placebo dose B every 2 weeks for a total of 3 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABBV-8736 — Intravenous (IV) Infusion
  Arms: Group 1: Dose A of ABBV-8736; Group 2: Dose B of ABBV-8736
Drug: Placebo — IV Infusion
  Arms: Group 1: Dose A of ABBV-8736 Placebo; Group 2: Dose B of ABBV-8736 Placebo

SUMMARY:
The objective of this study is to assess the safety, tolerability, pharmacokinetics, and immunogenicity following multiple intravenous (IV) ascending doses of ABBV-8736 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) is >= 18.0 to <= 32.0 kg/m^2 after rounding to the tenths decimal at Screening. BMI is calculated as weight in kg divided by the square of height measured in meters.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG.

Exclusion Criteria:

* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma as a child), renal, hepatic, gastrointestinal, hematologic or psychiatric disease or disorder, or any uncontrolled medical illness.
* History of any clinically significant sensitivity or allergy to any medication or food.
* Prior exposure to a TREM1 agent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to Approximately 113 Days
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Maximum Observed Concentration (Cmax) of ABBV-8736 | Up to Approximately 113 Days
  Cmax of ABBV-8736.
Time to Cmax (Tmax) of ABBV-8736 | Up to Approximately 113 Days
  Tmax of ABBV-8736.
Area under the plasma concentration-time curve from time 0 until the last measurable concentration (AUCtau) of ABBV-8736 | Up to Approximately 113 Days
  AUCtau of ABBV-8736.
Observed plasma concentration at the end of a dosing interval (Ctrough) of ABBV-8736 | Up to Approximately 113 Days
  Ctrough of ABBV-8736.
Apparent Terminal Phase Elimination Rate Constant (β) of ABBV-8736 | Up to Approximately 113 Days
  β of ABBV-8736.
Terminal Phase Elimination Half-Life (t1/2) of ABBV-8736 | Up to Approximately 113 Days
  t1/2 of ABBV-8736.
Clearance (CL) for Intravenous (IV) Dosing | Up to Approximately 113 Days
  CL for IV dosing.
Immunogenicity of ABBV-8736 as Determined by Anti-Drug Antibodies (ADAs) | Up to Approximately 113 Days
  Incidence and concentrations of ADAs. Neutralizing ADAs (NAb) may be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Acpru /Id# 277377, Grayslake, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-918